CLINICAL TRIAL: NCT02348385
Title: Imaging Extrastriatal Dopamine Release in Tobacco Smokers and Nonsmokers
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1106008678; 1K02DA031750-01A1 (NIH)
Record Dates: First submitted 2015-01-21; First posted 2015-01-28 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Nicotine Dependence
Keywords: amphetamine; cigarette smokers
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Amphetamine; Dextroamphetamine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples will be obtained for hormones and amphetamine drug levels
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy Tobacco Smokers: There is only one arm to the study. All subjects will receive amphetamine
  Interventions: Drug: Amphetamine
- Healthy Nonsmokers: There is only one arm to the study. All subjects will receive amphetamine
  Interventions: Drug: Amphetamine

INTERVENTIONS:
Drug: Amphetamine — Subjects will have 2 PET scans on the same day. Up to 3 hours before the second PET Scan, amphetamine (0.4mg/kg, orally) will be administered.
  Other Names: dextroamphetamine

SUMMARY:
The goal is to examine sex differences in amphetamine-induced dopamine release in tobacco smokers and nonsmokers.

DETAILED DESCRIPTION:
Aim 1:

To determine sex differences in amphetamine-induced dopamine (DA) release in healthy tobacco smokers and nonsmokers.

FLB-457 has been used in several PET centers and has recently been approved for use at the Yale University PET Center. We would like to determine whether there are sex differences in amphetamine induced DA release in healthy tobacco smokers and nonsmokers. Specifically, 40 healthy tobacco smokers and 40 healthy nonsmokers will have an magnetic resonance imaging (MRI) scan followed on another day by two FLB scans (ideally, the two PET scans will be carried out in the same day). Starting at 3 hours before the second PET scan, amphetamine (0.4mg/kg, PO) will be administered.

Aim 2:

To determine sex differences in amphetamine-induced dopamine release in tobacco smokers from Aim 1 after treatment with guanfacine. Guanfacine will be given under a different protocol. We plan to determine whether guanfacine treatment differentially inhibits amphetamine-induced DA release in men and smokers from Aim 1. After their first scan, the same 40 healthy tobacco smokers from Aim 1 will take guanfacine for 3 weeks under and then will have another set of FLB scans (ideally, the two PET scans will be carried out in the same day). Starting at 3 hours before the second PET scan, amphetamine (0.4mg/kg, PO) will be administered, as before. The sets of scans will be separated by at least 21 days, but due to scheduling and technical difficulties the second set may be scheduled up to 6 weeks after the first set.

ELIGIBILITY:
General inclusion criteria:

* men and women, aged 18-55 years
* who are able to read and write
* who are able to give voluntary written informed consent
* have no current uncontrolled medical condition such as neurological, cardiovascular, endocrine, renal, liver, or thyroid pathology
* have no history of a neurological or psychiatric disorder, e.g., no DSM-IV Axis 1 diagnosis in 2 preceding years)
* drink less than 21 drinks/week for women and less than 35 drinks per week for men
* have not used marijuana in the past 30 days and have not met criteria for dependence in the past 2 years
* do not suffer from claustrophobia or any MRI contradictions
* to participate in imaging studies including 2 PET scans and 1 MRI scan
* nonsmokers (smoked < 100 cigarettes in lifetime with urinary cotinine levels 0-30 ng/mL both at intake evaluation and on scan day)
* smokers (smoked at least 10 cigarettes/day for at least one year with an Fagerstrom score (FTND)>3, urine cotinine >150 ng/mL and carbon monoxide (CO) >12 ppm at intake)

General exclusion criteria:

* psychosis
* presence of acute or unstable medical or neurological illness. Subjects will be excluded from the study if they present with any history of serious medical or neurological illness or if they show signs of a major medical or neurological illness on examination or lab testing including history of seizures, head injury, brain tumor, heart, liver or kidney disease, eating disorder, diabetes.
* regular use of any psychotropic drugs including anxiolytics and antidepressants and other over-the-counter medications and herbal products within the last six months
* pregnancy/Breast feeding (as documented by pregnancy testing at screening or at days of the imaging studies),
* suicidal ideation or behavior
* pacemaker or other ferromagnetic material in body.
* use of medications which affect dopamine transmission within 2 weeks of the PET study
* Participation in other research studies involving ionizing radiation within one year of the PET scans that would cause the subject to exceed the yearly dose limits for normal volunteers.
* Blood donation within 8 weeks of the start of the study.
* history of a bleeding disorder or are taking medication to thin their blood

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Smokers and non smokers
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2012-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Cosgrove, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Tobacco Smokers | Healthy Nonsmokers
Started | 24 | 25
Completed | 24 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Tobacco Smokers: Healthy Tobacco Smoker Subjects will have 2 PET scans on the same day. Up to 3 hours before the second PET Scan, amphetamine (0.4mg/kg, orally) will be administered.
- Healthy Nonsmokers: Healthy Nonsmoker Subjects will have 2 PET scans on the same day. Up to 3 hours before the second PET Scan, amphetamine (0.4mg/kg, orally) will be administered.
- Total: Total of all reporting groups
Arm/Group | Healthy Tobacco Smokers | Healthy Nonsmokers | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 25 | 49
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 12 | 13 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 11 | 6 | 17
  White | 11 | 15 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Binding Potential of Dopamine Release During PET Scan Post Amphetamine Administration
Description: Percent change in binding potential of dopamine release during PET scan post amphetamine administration.Binding potential (BP) is the PET neuroimaging outcome measure that is computed as a proxy for availability of dopamine D2/3 receptors in a given region-of-interest.
Time Frame: After 2 PET Scans (1 day)
Measure: Mean (Standard Deviation); unit: percentage change in binding potential
Groups:
- Male Healthy Tobacco Smokers; Female Healthy Tobacco Smokers; Female Healthy Nonsmokers: Healthy Tobacco Smoker Subjects will have 2 PET scans on the same day. Up to 3 hours before the second PET Scan, amphetamine (0.4mg/kg, orally) will be administered.
- Male Healthy Nonsmokers: Healthy Nonsmoker Subjects will have 2 PET scans on the same day. Up to 3 hours before the second PET Scan, amphetamine (0.4mg/kg, orally) will be administered.
Arm/Group | Male Healthy Tobacco Smokers | Male Healthy Nonsmokers | Female Healthy Tobacco Smokers | Female Healthy Nonsmokers
Number analyzed (Participants) | 12 | 13 | 12 | 12
percentage change in binding potential | 14 (4.3) | 11.2 (2.4) | 1.9 (3.0) | 9.3 (3.3)

ADVERSE EVENTS:
Time Frame: Monitoring for adverse events was maintained from initial protocol approval to final subject participation, (5 years 4 months) Monitoring for each individual subject was maintained for at least one week after their final study visit or until any issues had resolved.
Description: No Reportable Adverse Events Occurred
Arm/Group | Healthy Tobacco Smokers | Healthy Nonsmokers
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 0/24 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT02348385/Prot_SAP_000.pdf